CLINICAL TRIAL: NCT05045846
Title: Diagnostic Accuracy of Rapid Antigen Test Based on Anterior Nasal Swab Compared With RT-PCR for SARS-CoV-2 Detection.
Status: Completed | Type: Observational
Sponsor: Christian von Buchwald (Other)
Responsible Party: Sponsor-Investigator, Christian von Buchwald, Medical Doctor, investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: COVID-19 rapid antigen test
Record Dates: First submitted 2021-09-14; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: rapid antigen test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to determine the accuracy of anterior nasal swab in rapid antigen (Ag)-tests in a low SARS-CoV-2 prevalence and massive screened community.

ELIGIBILITY:
Inclusion Criteria:

* Citizens, above 18 years of age, who had self-booked an appointment for COVID-19 test at Testcenter Taastrup, Copenhagen, Denmark, in the period of 2nd of March to 22nd of March were offered to participate in the project

Exclusion Criteria:

* Patients referred to COVID-19 testing by a doctor with symptoms of COVID-19 were tested in a separate section of the test centers and are not included in this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The infection pressure in the Capital Region of Denmark including Testcenter Taastrup was below 1.0%, throughout the study period
Sampling Method: Probability Sample
Enrollment: 3461 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of anterior nasal swab in rapid antigen (Ag)-tests | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Christian von Buchwald, MD, DMSc, Professor, Copenhagen, Denmark